CLINICAL TRIAL: NCT02639988
Title: Impact of Rheumatoid Arthritis on Type 2 Diabetes Mellitus
Brief Title: Impact of Rheumatoid Arthritis on the Course of Type 2 Diabetes During a Longitudinal Follow-up of 5 Years
Acronym: INSPIRED
Status: Terminated | Type: Observational
Why Stopped: Given the number of patients included in the cross-sectional analysis and the lack of financial resources, it was decided to focus on cross-sectional data.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI15005
Record Dates: First submitted 2015-11-30; First posted 2015-12-28 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes mellitus; Rheumatoid arthritis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- rheumatoid arthritis and type 2 diabetes
- osteoarthritis and type 2 diabetes

SUMMARY:
The purpose of this study is to determine whether patients with rheumatoid arthritis and type 2 diabetes experience a more severe disease course compared to control patients with osteoarthritis and type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

Patients

* Adults (>18 years)
* Rheumatoid arthritis fulfilling American College of Rheumatology (ACR )1987 or European League Against Rheumatism (ACR/EULAR) 2010 classification criteria
* Type 2 diabetes (HbA1c ≥6.5% OR fasting glycemia≥7 mmol/l OR glycemia 120 min after 75 mg glucose ingestion ≥ 11.1 mmol/l OR symptoms of hyperglycemia with glycemia ≥11.1 mmol/l)
* Affiliated to social security system

Controls

* Adults (>18 years) matched for age, sex and BMI with patients with rheumatoid arthritis
* Osteoarthritis (knee, hip, spine and hand)
* Type 2 diabetes with disease duration matched with patients with rheumatoid arthritis
* Affiliated to social security system

Exclusion Criteria:

* Patient not able to understand study implication and rules
* Patient opposed to participate to the study
* Transient diabetes
* Gestational diabetes
* Secondary diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients recruited in five rheumatology departments
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Time to the addition of a new treatment for type 2 diabetes in months | five years
  addition of a new treatment includes insulin requirement

SECONDARY OUTCOMES:
Glycated haemoglobin (HbA1c) levels in % | two years
Insulin resistance (HOMA-IR), absolute value | two years
Proportion of patients requesting insulin in % | two years
Proportion of patients with type 2 diabetes-related acute complications in % | two years
Proportion of patients requiring the addition of a new treatment for type 2 diabetes in % | five years
Proportion of patients with increased glycated haemoglobin (HbA1c) levels between 2 visits in % | five years
Proportion of patients with increased HOMA-IR between 2 visits in % | five years

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Avouac, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Cochin hospital, Paris, Paris, France

REFERENCES:
- [Background] Meune C, Touze E, Trinquart L, Allanore Y. High risk of clinical cardiovascular events in rheumatoid arthritis: Levels of associations of myocardial infarction and stroke through a systematic review and meta-analysis. Arch Cardiovasc Dis. 2010 Apr;103(4):253-61. doi: 10.1016/j.acvd.2010.03.007. Epub 2010 May 18. PMID 20656636
- [Background] Meune C, Touze E, Trinquart L, Allanore Y. Trends in cardiovascular mortality in patients with rheumatoid arthritis over 50 years: a systematic review and meta-analysis of cohort studies. Rheumatology (Oxford). 2009 Oct;48(10):1309-13. doi: 10.1093/rheumatology/kep252. Epub 2009 Aug 20. PMID 19696061
- [Background] Liao KP, Solomon DH. Traditional cardiovascular risk factors, inflammation and cardiovascular risk in rheumatoid arthritis. Rheumatology (Oxford). 2013 Jan;52(1):45-52. doi: 10.1093/rheumatology/kes243. Epub 2012 Sep 16. PMID 22986289
- [Background] Reilly MP, Wolfe ML, Rhodes T, Girman C, Mehta N, Rader DJ. Measures of insulin resistance add incremental value to the clinical diagnosis of metabolic syndrome in association with coronary atherosclerosis. Circulation. 2004 Aug 17;110(7):803-9. doi: 10.1161/01.CIR.0000138740.84883.9C. Epub 2004 Aug 2. PMID 15289378
- [Background] Chung CP, Oeser A, Solus JF, Gebretsadik T, Shintani A, Avalos I, Sokka T, Raggi P, Pincus T, Stein CM. Inflammation-associated insulin resistance: differential effects in rheumatoid arthritis and systemic lupus erythematosus define potential mechanisms. Arthritis Rheum. 2008 Jul;58(7):2105-12. doi: 10.1002/art.23600. PMID 18576352
- [Background] Dessein PH, Joffe BI. Insulin resistance and impaired beta cell function in rheumatoid arthritis. Arthritis Rheum. 2006 Sep;54(9):2765-75. doi: 10.1002/art.22053. PMID 16947779
- [Background] Ashida R, Ihn H, Mimura Y, Jinnin M, Asano Y, Kubo M, Tamaki K. Clinical features of scleroderma patients with contracture of phalanges. Clin Rheumatol. 2007 Aug;26(8):1275-7. doi: 10.1007/s10067-006-0490-0. Epub 2006 Dec 15. PMID 17171315
- [Background] Kiortsis DN, Mavridis AK, Vasakos S, Nikas SN, Drosos AA. Effects of infliximab treatment on insulin resistance in patients with rheumatoid arthritis and ankylosing spondylitis. Ann Rheum Dis. 2005 May;64(5):765-6. doi: 10.1136/ard.2004.026534. Epub 2004 Sep 30. PMID 15458960
- [Background] Rosenvinge A, Krogh-Madsen R, Baslund B, Pedersen BK. Insulin resistance in patients with rheumatoid arthritis: effect of anti-TNFalpha therapy. Scand J Rheumatol. 2007 Mar-Apr;36(2):91-6. doi: 10.1080/03009740601179605. PMID 17476613
- [Background] Solomon DH, Massarotti E, Garg R, Liu J, Canning C, Schneeweiss S. Association between disease-modifying antirheumatic drugs and diabetes risk in patients with rheumatoid arthritis and psoriasis. JAMA. 2011 Jun 22;305(24):2525-31. doi: 10.1001/jama.2011.878. PMID 21693740
- [Background] Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006 Dec 7;355(23):2427-43. doi: 10.1056/NEJMoa066224. Epub 2006 Dec 4. PMID 17145742
- [Background] Arrieta F, Pinera M, Iglesias P, Nogales P, Salinero-Fort MA, Abanades JC, Botella-Carretero JI, Calanas A, Balsa JA, Zamarron I, Rovira A, Vazquez C; ESD2 Group. Metabolic control and chronic complications during a 3-year follow-up period in a cohort of type 2 diabetic patients attended in primary care in the Community of Madrid (Spain). Endocrinol Nutr. 2014 Jan;61(1):11-7. doi: 10.1016/j.endonu.2013.09.002. Epub 2013 Oct 30. PMID 24182687